CLINICAL TRIAL: NCT06310187
Title: Oxidative Stress and Harmful Constituent Levels Associated With Little Cigars
Brief Title: Little Cigar Oxidants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joshua Muscat, Professor, Department of Public Health Sciences, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY000023967; U54DA058271-01 (NIH)
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use; Oxidative Stress
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Williams Design for Cross over-trials with a 3-period 3-treatment cross-over design in 36 healthy daily cigarette smokers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Subjects will be given the high oxidant little cigar for their first laboratory visit. They will then be given the low oxidant little cigar for the second visit followed by using their own cigarette at the final laboratory visit.
  Interventions: Other: High Oxidant Little Cigar; Other: Low Oxidant Little Cigar; Other: Usual Cigarette
- Group B (Experimental): Subjects will be given the low oxidant little cigar for their first laboratory visit. They will then use their own cigarette for the second visit followed by being given the high oxidant little cigar at the final laboratory visit.
  Interventions: Other: High Oxidant Little Cigar; Other: Low Oxidant Little Cigar; Other: Usual Cigarette
- Group C (Experimental): Subjects will use their own cigarette for their first laboratory visit. They will then be given the high oxidant little cigar for the second visit followed by being given the low oxidant little cigar at the final laboratory visit.
  Interventions: Other: High Oxidant Little Cigar; Other: Low Oxidant Little Cigar; Other: Usual Cigarette

INTERVENTIONS:
Other: High Oxidant Little Cigar — Subjects will be given a high oxidant little cigar to use for outcome measure data collection in the lab before and after product usage.
Other: Low Oxidant Little Cigar — Subjects will be given a low oxidant little cigar to use for outcome measure data collection in the lab before and after product usage.
Other: Usual Cigarette — Subjects will use their own cigarette for outcome measure data collection in the lab before and after product usage.

SUMMARY:
Determine the effects of little cigars on human exposure to tobacco smoke oxidants. In a balanced randomized cross-over study design in cigarette smokers, subjects will be assigned to 3 exposure groups. These include a high oxidant little cigar exposure condition, a low oxidant little cigar exposure condition, and their usual cigarette. Biological samples will be collected before and after product usage.

DETAILED DESCRIPTION:
Exhaled breath condensate samples will be collected at pre-product usage, post-product usage, 30, and 60 minutes. Samples will be analyzed for levels of oxidant markers including 8-isoprostanes, 8-OHdG acrolein adducts and C-reactive protein.

Exhaled breath samples will be collected at pre-product usage and post-product usage. Samples will be analyzed for levels of oxidant markers in Volitive Organic Compound (VOC) profiles.

Blood samples will be collected at pre-product usage and post-product usage. Samples will be analyzed nicotine, 8-isoprostane and other oxidative makers of stress.

Buccal cell samples will be collected at pre-product usage and post-product usage. Samples will be analyzed for 8-OHdG adducts.

Salvia samples will be collected at pre-product usage and post-product usage. Samples will be analyzed for 8-OHdG adducts and metabolomic profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 - 65 years old
2. Daily cigarette smoker (>= 1 cigarette per day);
3. Smoke regular, filtered cigarettes or machine rolled cigarettes with a filter
4. No current or past use of Little Cigars
5. All other forms of nicotine must be used <6 days out of the past 30 days.
6. Able to read and write in English
7. No serious cigarette smoking quit attempt or use of any FDA-approved smoking cessation medication in the prior 30 days
8. No plan to quitting smoking in the next 3 months

Exclusion Criteria:

1. Women who are pregnant and/or nursing or trying to become pregnant
2. Unstable or significant medical condition in the past 3 months (e.g., recent heart attack or other serious heart condition, stroke, severe angina)
3. Respiratory diseases (e.g., exacerbations of asthma or Chronic Obstructive Pulmonary Disease (COPD), require oxygen, require oral prednisone), kidney (e.g., dialysis) or liver disease (e.g., cirrhosis), severe immune system disorders (e.g., uncontrolled HIV/AIDS, multiple sclerosis symptoms) or any medical disorder/medication that may affect participant safety or biomarker data
4. Uncontrolled substance abuse or inpatient treatment for that condition in the past 6 months
5. Exhaled Carbon Monoxide (CO) measurement of >= 17 parts per million

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
8-isoprostanes Concentration in Exhaled Breath Condensate | -5 minutes
8-OHdg Acrolein Adduct Concentration in Exhaled Breath Condensate | -5 minutes
C-reactive Protein Concentration in Exhaled Breath Condensate | -5 minutes
8-isoprostanes Concentration in Exhaled Breath Condensate | 0 minutes
8-OHdg Acrolein Adduct Concentration in Exhaled Breath Condensate | 0 minutes
C-reactive Protein Concentration in Exhaled Breath Condensate | 0 minutes
8-isoprostanes Concentration in Exhaled Breath Condensate | 30 minutes
8-OHdg Acrolein Adduct Concentration in Exhaled Breath Condensate | 30 minutes
C-reactive Protein Concentration in Exhaled Breath Condensate | 30 minutes
8-isoprostanes Concentration in Exhaled Breath Condensate | 60 minutes
8-OHdg Acrolein Adduct Concentration in Exhaled Breath Condensate | 60 minutes
C-reactive Protein Concentration in Exhaled Breath Condensate | 60 minutes
Oxidant makers in Volitive Organic Compound Profiles in Exhaled Breath Samples | -5 minutes
Oxidant makers in Volitive Organic Compound Profiles in Exhaled Breath Samples | 0 minutes
Nicotine concentration in Blood Samples | -5 minutes
Nicotine concentration in Blood Samples | 0 minutes
8-isoprostanes Concentration in Blood Samples | -5 minutes
8-isoprostanes Concentration in Blood Samples | 0 minutes
8-OHdg Acrolein Adduct Concentration in Buccal Cell Samples | -5 minutes
8-OHdg Acrolein Adduct Concentration in Buccal Cell Samples | 0 minutes
8-OHdg Acrolein Adduct Concentration in Saliva Samples | -5 minutes
8-OHdg Acrolein Adduct Concentration in Saliva Samples | 0 minutes
Metabolomic Profiles in Saliva Samples | -5 minutes
Metabolomic Profiles in Saliva Samples | 0 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Muscat, Ph.D., Principal Investigator — Penn State Hershey College of Medicine

IPD SHARING:
Plan to Share IPD: No